CLINICAL TRIAL: NCT01798446
Title: A Phase II Study of Axitinib in Metastatic Non-clear Cell Renal Cell Carcinoma Patients Previously Treated With Temsirolimus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Se-Hoon Lee, Associate Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-1301-124-461; SNUH_Axitinib_NCCRCC (Other: SNUH)
Record Dates: First submitted 2013-02-20; First posted 2013-02-25 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Renal Cell Carcinoma; Nonclear Cell; Temsirolimus Resistance
Keywords: Renal cell carcinoma; Nonclear cell; Temsirolimus resistance
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Axitinib (Experimental): This is a single arm study. Axitinib arm is the only arm who receive axitinib.
  Interventions: Drug: Axitinib

INTERVENTIONS:
Drug: Axitinib — Axitinib 5mg twice will be orally administered daily with one cycle of 4 weeks. The package of axitinib must be opened right before the administration due to its photosensitivity.

SUMMARY:
* 1. There is no standard treatment option for non-clear cell renal cell carcinoma (RCC).
* 2. Patients with non-clear cell RCC is strongly assumed to have benefit from anti-VEGF treatment.
* 3. There is no trial of axitinib for non-clear cell RCC.
* 4. Axitinib is expected to show more potent efficacy over sorafenib or sunitinib in renal cell carcinoma.

DETAILED DESCRIPTION:
1. Renal Cell Carcinoma Renal cell carcinoma is a malignant tumor occurring most frequently of primary malignant tumors in kidney.1 According to Korea Central Cancer Registry (KCCR) data, renal cancer affects 4.4 out of 100,000 males and 2.1 out of 100,000 females. About 30% of renal cancer patients accompany remote metastasis at the time of diagnosis and renal cancer even recurs in about 40% of the patients who underwent surgery for radical treatment of renal cancer as a local disease.1 New treatment strategies against renal cell carcinoma have been developed, but they have not obtained satisfactory therapeutic outcomes. Thus, constant clinical studies are necessary to improve therapeutic efficacy.
2. Treatment of Metastatic Renal Cell Carcinoma The treatment for metastatic renal cell carcinoma has been improved a lot for the recent few years, which is, however, limited to clear cell renal cell carcinoma. The drugs showing antitumor activity against clear cell renal cell carcinoma include axitinib, sunitinib, sorafenib, bevacizumab, temsirolimus, and everolimus.

   Of them, axitinib, sunitinib, sorafenib, bevacizumab, etc. are neovascularization inhibitors which inhibit vascular endothelial growth factor (VEGF) and its receptor (VEGFR). As a first-line treatment, sunitinib prolongs progression-free survival (PFS) compared to interferon-alpha, being recognized as a first-line standard therapy. Sorafenib, a second-line treatment, shows significant prolongation of PFS against clear cell renal cell carcinoma compared to the placebo control group, establishing itself as a second-line drug. Concomitantly administered with interferon-alpha, bevacizumab shows significant prolongation of PFS compared to the single use of interferon-alpha, establishing itself as another first-line therapy. Temsirolimus, an mammalian target of rapamycin (mTOR) inhibitor, extended survival time in a clinical study of both clear and non-clear cell renal cell carcinoma. However, this clinical study was limited to patients with renal cell carcinoma having bad prognostic factors. This renal cell carcinoma with bad prognostic factors only accounts for 10-20% of entire metastatic renal cell carcinoma. Everolimus, an another mTOR inhibitor, showed a significant prolongation of PFS in the placebo-controlled phase III clinical study of patients with clear cell renal cell carcinoma in whom sunitinib therapy failed, establishing itself as a second-line therapy in case the first-line standard sunitinib therapy fails.
3. Treatment of Metastatic Non-clear Cell Renal Cell Carcinoma (nccRCC) In fact, VEGF antagonists are shown to have some efficacy also in nccRCC. Sunitinib was effective against nccRCC. A worldwide expanded access trial of sunitinib has been undertaken. A subgroup analysis of patients with non-clear-cell histology was performed and 276 patients (11.8%) with non-clear-cell histology were identified, although distinction between different subtypes was not made. A response rate of 5.4%, clinical benefit (defined as response and stable disease was more than 3 months) of 47% and median PFS of 6.7 months was seen in this subgroup. This result compared with an overall response rate for the entire patient group of 9.3%, clinical benefit of 52.3%, and median PFS of 8.9 months. The investigators concluded that sunitinib was active in the non-clear-cell subgroup; however, these data need to be interpreted with caution because of the nonrandomization of patients in the expanded access trial and the lack of pathology verification. Also, recently, phase 2 trial of sunitinib in non-clear cell renal cell carcinoma showed remarkable efficacy with response rate of 36% and median PFS of 6.4 months. The study enrolled non-clear cell RCC patients who did not receive previous anti-angiogenic treatment.

   Sorafenib also showed some efficacy in nccRCC, though not so efficacious. The Advanced Renal Cell Carcinoma Sorafenib Expanded Access Program allowed patients in the United States and Canada with metastatic RCC to receive treatment with sorafenib prior to its regulatory approval. This non-randomized, open-label program treated 158 subjects with papillary RCC of a total of 1891 evaluable subjects (81% clear cell, 8% non-clear, and 11% unclassified histology). Of the 107 evaluable subjects with papillary RCC, 90 (84%) had a measurable response to treatment with 3 partial responders and 87 with stable disease for at least 8 weeks, while 17 (16%) subjects demonstrated early progression on treatment. The side effect profile for sorafenib was similar across histologic subtypes, and the authors concluded that sorafenib has some activity in papillary tumors.

   On the other hand, in randomized phase 3 trial of single-agent Axitinib in 723 renal cell carcinoma patients who progressed despite first-line therapy containing sunitinib, bevacizumab plus interferon-alpha, temsirolimus or cytokines, the median PFS duration was significantly longer with axitinib than with sorafenib in the entire population (6.7 months versus 4.7 months, respectively: p less than 0.0001).
4. Rationale In short,

   1. There is no standard treatment option for non-clear cell RCC.
   2. Patients with non-clear cell RCC is strongly assumed to have benefit from anti-VEGF treatment.
   3. There is no trial of axitinib for non-clear cell RCC.
   4. Axitinib is expected to show more potent efficacy over sorafenib or sunitinib in renal cell carcinoma.

Based on above, this clinical study is designed to examine efficacy and adverse events of axitinib for non-clear cell renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmation of RCC without a clear cell histologic component, e.g., papillary type, chromophobe type, medullary type or unclassified)
* Patients with stage IV or recurrent disease not amenable to surgery, radiotherapy, or combined modality therapy with curative intent
* Previous treatment with temsirolimus
* Measurable disease according to RECIST criteria
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Age 18 years or older
* Adequate cardiac function
* Adequate bone marrow, hepatic, and renal function
* Hematology:

Neutrophil same or more than 1.5 x 10^9/L Platelet same or more than 75 x 10^9/L Hemoglobin same or more than 9 g/dL -Liver function tests: Total bilirubin same or less than 1.5 x upper limit normal (xULN) aspartate aminotransferase(AST), alanine aminotransferase (ALT) same or less than 2.5 xULN Alkaline phosphatase same or less than 2.5 xULN

-Renal function tests: Creatinine clearance same or more than 30 mL/min

* Life expectancy more than 3 months
* Signed and dated informed consent of document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment

Exclusion Criteria:

* Clear cell type RCC
* Composed of mostly sarcomatoid carcinoma
* Collecting duct type RCC
* Diagnosis of any serious secondary malignancy within the last 2 years, except for adequately treated basal cell or squamous cell carcinoma of skin, or in situ carcinoma of cervix uteri
* Hypertension that cannot be controlled by medications (blood pressure 150/90 mmHg despite optimal medical therapy)
* Pregnancy or breast feeding
* Other severe acute or chronic medical or psychiatric condition
* Prior treatment on sunitinib, sorafenib, pazopanib or bevacizumab
* Uncontrolled central nerve system (CNS) metastasis (brain and/or leptomeningeal metastasis)
* Patients who require concomitant treatment with potent cytochrome P 3A4 ( CYP3A4) inducers and inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-02; Primary Completion 2015-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | Followed up during study drug administration till disease progression, unacceptable toxicitiy, or 1 year
  PFS is a time from study enrollment to documented disease progression or death from any cause

SECONDARY OUTCOMES:
Response Rate | Every 8 weeks till disease progression, unacceptable toxicity or 1 year
  Tumor response according to Response Evaluation Criteria for Solid Tumor (RECIST) criteria version 1.1
Disease control rate (DCR) | Every 8 weeks till disease progression, unacceptable toxicity or 1 year
  Disease control (complete remission + partial remission + stable disease) rate according to RECIST criteria version 1.1
Overall survival | Every 8 weeks till disease progression, unacceptable toxicity or 1 year
  Duration from study enrollment to death from any cause
Number of patients who experience adverse events related to drug and serious adverse events | Every 4 weeks till disease progression, unacceptable toxicity or 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Se-Hoon Lee, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seou National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Rini BI, Escudier B, Tomczak P, Kaprin A, Szczylik C, Hutson TE, Michaelson MD, Gorbunova VA, Gore ME, Rusakov IG, Negrier S, Ou YC, Castellano D, Lim HY, Uemura H, Tarazi J, Cella D, Chen C, Rosbrook B, Kim S, Motzer RJ. Comparative effectiveness of axitinib versus sorafenib in advanced renal cell carcinoma (AXIS): a randomised phase 3 trial. Lancet. 2011 Dec 3;378(9807):1931-9. doi: 10.1016/S0140-6736(11)61613-9. Epub 2011 Nov 4. PMID 22056247
- See also: Related Info — http://hmo.snuh.org/